CLINICAL TRIAL: NCT06058351
Title: ABI-aftercare in Motion: Multidisciplinary Aftercare in the Home Environment in Patients With Acquired Brain Injury; an Implementation Study
Brief Title: ABI-aftercare in Motion: Multidisciplinary Aftercare in the Home Environment in Patients With Acquired Brain Injury
Acronym: ABI-motion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Majanka H. Heijenbrok-Kal, PhD (Other)
Collaborators: Netherlands Brain Foundation (Other)
Responsible Party: Sponsor-Investigator, Majanka H. Heijenbrok-Kal, PhD, Clinical epidemiologist, Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 11172
Record Dates: First submitted 2023-09-08; First posted 2023-09-28 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Acquired Brain Injury
Keywords: Acquired Brain Injury; Rehabilitation; Aftercare; Implementation
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Intervention Model Description: A group of patients will be followed during standard outpatient rehabilitation before and after implementation of the ABI-motion program with 1 year follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ABI-motion group (Experimental): Patients following outpatient rehabilitation after implementation of the ABI-motion program
  Interventions: Behavioral: ABI-motion program
- Control group (No Intervention): Patients following outpatient rehabilitation before implementation of the ABI-motion program

INTERVENTIONS:
Behavioral: ABI-motion program — The ABI-motion program strengthens the cooperation between outpatient rehabilitation professionals and community care providers.
  Arms: ABI-motion group

SUMMARY:
The goal of this implementation study is to improve aftercare for patients with ABI receiving outpatient rehabilitation. The ABI-motion program was developed to improve and active lifestyle and to prevent persistent complaints after ABI and poor HR-QoL.The main questions it aims to answer are:

* Is the ABI-motion program feasible?
* What are the health benefits of the ABI-motion program?

Participants will receive brain education, a joint therapy session with a physical or occupational or movement therapist and a buddy from a patient support organization during outpatient rehabilitation, followed by community buddy support after discharge from outpatient rehabilitation, and follow-up by a rehabilitation physician.

DETAILED DESCRIPTION:
Rationale: Many people with acquired brain injury (ABI) experience difficulties in reintegration into their social life after discharge from the rehabilitation center. It is also known that people with ABI do not meet the physical activity guidelines; they have lower physical activity levels than healthy people and they have difficulty maintaining their physical fitness level reached during rehabilitation. An inactive lifestyle may lead to persistent complaints, such as fatigue, anxiety or depression, and may result in a poor health-related quality of life (HR-QoL).

Objective: To improve aftercare for patients with ABI receiving outpatient rehabilitation, aimed at promoting an active lifestyle to prevent persistent complaints after ABI and poor HR-QoL.

Study design: Care improvement study using a prospective mono-center cohort with a pre-post implementation study design.

Study population: Patients with ABI receiving outpatient rehabilitation therapy.

Intervention (if applicable): Implementation of an aftercare program that strengthens the cooperation between rehabilitation center and local patient support organisations in the community. The aftercare program integrates standard outpatient rehabilitation and community services, including: 1) brain education regarding long-term consequences of ABI, physical activity guidelines, and patient support organizations in the area; 2) a joint physical/ occupational/ movement therapy session with a buddy from a patient support organisation during outpatient rehabilitation; 3) buddy support (max 8 hrs) in the community towards an active lifestyle after rehabilitation discharge; 4) follow-up by the rehabilitation physician.

Main study parameters/endpoints: The proportion of participants with ABI participating in the community buddy program (target 60%) and feasibility (rating of satisfaction) of the program will be calculated. Secondary, objectively measured physical activity, physical fitness and cognitive functioning and patient reported outcomes (physical activity, fatigue, anxiety, depression, cognitive complaints, coping, community integration, HRQoL, physical fitness, health care use, return to work) using validated questionnaires will be collected before and at 3, 6, and 12 months after outpatient rehabilitation discharge.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ABI
* Follows an outpatient rehabilitation program for ABI in Rijndam Rehabilitation

Exclusion Criteria:

* Having a contra-indication for participation in moderate to vigorous exercise
* Life expectancy < 1 year
* Incapacitated persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Difference in proportion of patients participating in buddy support programs after rehabilitation discharge | 3, 6, 12 months
  Proportion of patients in the ABI-motion group that continues community buddy support after rehabilitation discharge compared with standard care
Mean rating of satisfaction with the ABI-motion program | 12 months
  Satisfaction with the ABI-motion program is rated on a rating scale, ranging from 0 (worst) to 10 (best).

SECONDARY OUTCOMES:
Change in total minutes of physical activity/week at 6 and 12 months compared with controls | 0, 6, 12 months
  Physical activity is measured with an activity monitor (min/week) and electronic diary
Change in Montreal Cognitive Assessment (MoCA) score at 6 and 12 months compared with controls. | 0, 6,12 months
  The MoCA is a screening tool for detection of mild cognitive impairment. The total score ranges from 0 (worst) to 30 (best).
Change in functional exercise capacity at 6 and 12 months compared with controls | 0, 6, 12 months
  The 1-minute Sit-to-Stand Test (1mSTS) measures the number of sit-to-stand transitions during 1 minute.
Change in Walking Speed at 6 and 12 months compared with controls | 0, 6, 12 months
  10 meter Walk Test (10mWT) assesses walking speed (m/s) over a short duration.
Change in handgrip strength at 6 and 12 months compared with controls | 0, 6, 12 months
  Maximum isometric handgrip strength is measured with a hand-held dynamometer over 6 attempts (3 per hand) in kg.
Change in anxiety and depression at 3, 6, and 12 months compared with controls | 0, 3, 6, and 12 months
  The Hospital Anxiety and Depression Scale (HADS) subscale scores are used to measure Anxiety and Depression, 7 items each, with subscale scores ranging from 0 (best) to 21 (worst), with scores 0-7 indicating normal sores, 8-10 borderline cases, and 11-21 definite cases of anxiety or depression.
Change in fatigue at 3, 6, and 12 months compared with controls | 0, 3, 6, and 12 months
  The Checklist Individual Strength (CIS) consists of 20 statements on fatigue-related problems respondents might have experienced in the past 2 weeks. The items are rated on a 1-7 point Likert scale, with total scores ranging from 20 (best) to 140 (worst).
Change in cognitive failures at 3, 6, and 12 months compared with controls | 0, 3, 6, and 12 months
  The Cognitive Failures Questionnaire (CFQ) is used to assess the frequency with which people experience cognitive failures in everyday life, such as absent-mindedness, slips and errors of perception, memory, and motor functioning. The total score of the scale is the sum of the ratings of the 25 individual items, yielding a score from 0 (best) to 100 (worst).
Change in coping style at 3, 6, and 12 months compared with controls | 0, 3, 6, and 12 months
  The short version of the Coping Inventory for Stressful Situations (CISS-SF) is used as a measure of coping with stressful situations. It has 21 items which are rated on a 1(no) to 5 (strong) point rating scale. It contains 3 subscales: task-oriented, emotion-oriented, and avoidance-oriented coping. Each subscale score ranges from 7 (low use) to 35 (high use), with higher scores indicating a greater use of that particular coping strategy.
Change in health-related quality of life at 3, 6, and 12 months compared with controls | 0, 3, 6, 12 months
  The EQ-5D-5L consists of the 5-item EQ-5D index (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) and a visual analogue scale (EQ VAS). The 5 EQ-5D index items are summarized into a weighted overall score, which runs from 0 for the value of death to 1.00 for full health. The EQ VAS ranges from 0 to 100 (worst to best imaginable health state).
Change in physical and mental components of health-related quality of life at 3, 6, and 12 months compared with controls | 0, 3, 6, 12 months
  The Short Form-36 contains 36 items measuring multidimensional quality of life. A physical component summary (PCS) and a mental component summary (MCS) can be calculated, which are T-scores, having a mean of 50 and standard deviation of 10.
Change in physical activity at 3, 6,12 months compared with controls | 0, 3, 6, 12 months
  The International Physical Activity Questionnaire assesses the time spent (min. per week) in several types of physical activity (vigorous activities, moderate activities, walking, and sitting) that people do as part of their daily lives.
Change in fitness at 3, 6,12 months compared with controls | 0, 3, 6, 12 months
  The International Fitness Scale (IFIS) questionnaire gives a measure of fitness based on the answers to 5 basic questions about fitness: physical fitness, cardiorespiratory fitness, muscular fitness, speed-agility, flexibility, and overall fitness, with answers based on a 5-point Likert-scale (1=very poor, to 5=very good).
Change in social participation and health care use at 3, 6, 12 months compared with controls | 0, 3, 6, 12 months
  The Utrecht Scale for Evaluation of Rehabilitation - Participation (USER-P) contains 32 questions with three scales measuring the frequency of participation, perceived participation restrictions, and satisfaction with participation in society. Total scores range from 0 (worst) to 100 (best).
Change in health care use at 3, 6, 12 months compared with controls | 0, 3, 6, 12 months
  The iMTA Medical Consumption Questionnaire is an instrument to measure medical consumption. It includes questions related to the frequency of contacts with health care providers.
Change in medical consumption at 3, 6, 12 months compared with controls | 0, 3, 6, 12 months
  The iMTA Productivity Cost Questionnaire (iPCQ) is used to measure the costs (Dollars and/or Euros) of productivity losses.

CONTACTS AND LOCATIONS:
Overall Officials: Gerard M Ribbers, MD, PhD, Study Chair — Erasmus Medical Center
Locations (1):
- Rijndam Rehabilitation, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
upon request
Supporting Information: Study Protocol, SAP, ICF